CLINICAL TRIAL: NCT00305331
Title: Phase II Clinical Trial of Domperidone as a Treatment for Dopamine Agonist-induced Peripheral Edema in Patients With Parkinson's Disease
Brief Title: Domperidone as a Treatment for Dopamine Agonist-induced Peripheral Edema in Patients With Parkinson's Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of recruitment
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Susan Fox, PI, University Health Network, Toronto
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: MDCDOM2006
Record Dates: First submitted 2006-03-20; First posted 2006-03-21 (Estimated); Last update posted 2012-07-30 (Estimated); Status verified 2012-07

CONDITIONS: Parkinson's Disease; Peripheral Edema
Keywords: Parkinson's disease; Domperidone; Peripheral edema; Pramipexole; Ropinirole
MeSH Terms: conditions — Parkinson Disease | interventions — Domperidone; Pharmaceutical Preparations

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

INTERVENTIONS:
Drug: Domperidone (drug)

SUMMARY:
The dopamine agonists, pramipexole (Mirapex) and ropinirole (Requip), are drugs that are used to treat symptoms of Parkinson's disease. However, these drugs can induce bothersome leg swelling or edema in about 20 percent of patients. The cause of this edema is unknown but may be secondary to stimulation of peripheral dopamine receptors in the kidney or blood vessels. We hypothesise that a peripherally acting dopamine receptor antagonist, will reduce edema in PD patients. This study will assess the effect of the peripheral acting dopamine D2 receptor antagonist, domperidone as a potential treatment for dopamine agonist-induced leg swelling.

DETAILED DESCRIPTION:
The study is a phase II, randomised double-blind, placebo-controlled, cross-over trial. There are four periods: recruitment and randomisation; treatment period one (4 weeks); washout (1 week); and finally treatment period two (4 weeks). Patients will be randomly assigned domperidone 20 mg tid in treatment period one followed by placebo tid in treatment period two, or placebo tid in treatment period one followed by domperidone 20 mg tid in treatment period two.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic PD
* On a stable medication regimen for at least one month with leg edema occurring after the start of pramipexole or ropinirole and the absence of other possible reasons for discontinuation of pramipexole or ropinirole treatment (e.g. other adverse effects).

Exclusion Criteria:

* Pregnancy
* Breastfeeding
* Women of child bearing age not using a reliable method of contraception
* Coronary disease, abnormal QT interval on electrocardiogram (EKG)
* Diabetes mellitus
* Hepatic disease
* Alcohol abuse
* Renal disease
* Edema of one leg only
* Presence of other conditions possibly causing leg edema

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2006-03; Primary Completion 2008-07 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
left foot volume measured by water displacement

SECONDARY OUTCOMES:
subjective reporting of leg oedema; UPDRS, CGI and adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Susan H Fox, Principal Investigator — Toronto Western Hospital, UHN
Locations (1):
- Movement Disorders Clinic, Toronto Western Hospital, 399, Bathurst St, Toronto, Ontario, Canada